CLINICAL TRIAL: NCT04040660
Title: Use of NexoBrid for Treatment of Acute Deep Partial and Full Thickness Burn Injuries
Acronym: NEXT
Status: Approved for marketing | Type: Expanded Access
Sponsor: MediWound Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MW2018-06-21
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Thermal Burn

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: NexoBrid — NexoBrid is presented as lyophilized powder and gel vehicle for preparation of a gel for cutaneous use. The API is a concentrate of proteolytic enzymes enriched in Bromelain extracted from the stem of Ananas comosus (pineapple plant)

SUMMARY:
Enzymatic eschar removal with NexoBrid allows initiating and completing the phase of removal of the offending eschar earlier upon admission, enabling earlier visualization of the wound bed for assessment of burn wound depth as well as preservation of viable dermal tissues, as further elaborated and supported by previous clinical studies. The depth determination is important for the planning and execution of the post eschar removal stage of wound closure phase (grafting or spontaneous epithelialization).

Additional clinically meaningful attributes of NexoBrid enzymatic eschar removal is the ability to lower surgical burden as it allows to remove eschar in wounds that otherwise would have to undergo surgical excision as no other non-surgical treatment is available for early and effective eschar removal.

MediWound has completed the recruitment of patients to study MW2010-03-02 (DETECT Study). The timeline for patients' follow-up and potential for approval in 2021/2022, creates a significant gap in the ability of clinical practitioner's to maintain their knowledge and skills in using NexoBrid as they no longer treat eligible patients. The expanded access protocol will allow to expand treatment to additional patients in up to 30 US burn centers (DETECT sites and additional sites). The proposed protocol will allow product availability to eligible population and keep the clinical use of the product knowledge active in the burn care community introducing it to their routine burn care.

The BLA assessment was completed and NexoBrid is approved for use in adults in the US. Adult enrollment is closed, and only pediatric patients will continue to be recruited for this treatment protocol.

The purpose of this treatment protocol is to provide NexoBrid to patients with DPT and FT thermal burns on up to 30% TBSA.

This protocol is also designed to collect and evaluate the safety and clinical performance of NexoBrid in this patient population.

DETAILED DESCRIPTION:
This is an Expanded Access (treatment) protocol to allow ongoing treatment of burn patients with NexoBrid following completion of the enrollment stage of protocol MW2010-03-02 (DETECT study).

This protocol is also designed to collect and evaluate the safety and clinical performance of NexoBrid in patients suffering from DPT and FT thermal burns.

Following the enrollment of a patient to the protocol, physicians will identify one or more target wounds (TWs) per patient according to the TW definition. All patient's DPT and FT burns that comply with the specified entrance criteria will be treated with NexoBrid and, therefore, must be designated as TWs. This will further allow an evaluation of the patient's systemic safety by allowing treatment of the patient's entire deep burns.

Prior to initiation of eschar removal treatment, patients will be medicated with appropriate analgesia and undergo wound cleansing and dressing of all wounds with antibacterial solutions according to product instruction for use in order to ensure clean and moist eschar covered wound bed for NexoBrid application. Vital signs (Blood Pressure, Heart Rate and temperature) measurements and pain assessment will be performed within 24 hrs before start of treatment as well as haematology, biochemistry blood tests & PTT/INR. Pressure measurements for circumferential extremity wounds will be performed 1 hour before start of treatment and will be closely monitored during treatment. Following wound cleansing and soaking treatments, patients will undergo the eschar removal process. TWs of up to 15% total body surface area (TBSA) will be treated with a single application of NexoBrid for 4 hours. Patients with TWs >15% TBSA and up to 30% TBSA will be treated with 2 consecutive applications of 4 hours each. NexoBrid should not be applied to more than 15% TBSA in one session. PK samples will be taken from sub-set of patients with TWs area >15% TBSA. Pressure measurements for circumferential extremity wounds will be performed after the removal of NexoBrid.

Post eschar removal completion, patients will undergo daily vital signs (Blood Pressure, Heart Rate and temperature measurements) and pain assessments for 1 week, starting on the morning following start of eschar removal. Blood tests (haematology and biochemistry) will be performed 24 ± 6 hrs post eschar removal as well as PTT/INR. Weekly assessments of wound healing progress including the dressings used until complete wound closure will be performed.

Cosmesis (scar quality) evaluation (using MVSS) will be performed at 3 and 12 months post wound closure confirmation visit.

ELIGIBILITY:
Inclusion Criteria patient level:

1. Pediatric only (0 to < 18years old) males and females
2. Thermal burns caused by fire/flame, scalds or contact,
3. Patient total burns area ≥ 1% DPT and / or FT with eschar that should be removed in SOC,
4. Patient total burns area to be treated should be ≤ 30% TBSA; SPT, DPT and/or FT in depth,
5. Informed consent can be obtained within 84h of the burn injury,
6. Patients and/or legal authorized representative who are willing and able to sign a written consent .

Inclusion Criteria - Wound level

* At least one wound (a continuous burn area) that is ≥0.5% TBSA (DPT and/or FT) (this minimal wound size should not include face, perineal or genital)

All planned TWs should meet the following criteria:

* SPT areas that cannot be demarcated from DPT and FT areas should be less than 50% of the % TBSA of the TW,
* Wound's blisters can be removed/ unroofed, as judged by the investigator.

Exclusion Criteria patient level:

1. Patients weighing less than 3kg,
2. Patients with burned, charred fingers, 3rd degree in depth and possibly devoid of circulation,
3. Patients with abraded wound/s that cannot be treated by an enzymatic debrider application (NexoBrid),
4. Patients with pre enrolment escharotomy,
5. Patients with electrical or chemical burns,
6. The following pre-enrollment dressings: a. Flammacerium, b. Silver Nitrate (AgNO3),
7. Patients with pre-enrolment wounds which are covered by eschar heavily saturated with Silver, Iodine or by SSD pseudoeschar (pseudoeschar as a result of > 12 hrs SSD treatment),
8. Patients with diagnosed infections as described in the protocol,
9. Diagnosis of smoke inhalation injury [12],
10. Pregnant women (serum positive pregnancy test) or nursing mothers,
11. Poorly controlled diabetes mellitus (HbA1c>11%) in patients with known diabetes as captured in the medical history,
12. BMI greater than 40.0 kg/m2,
13. American Society of Anesthesiologists (ASA) physical status classification system greater than 2
14. Cardio-pulmonary disease (MI within 6 months prior to injury, severe or unstable Ischemic Heart Disease, severe or unstable heart failure, severe pulmonary hypertension, severe COPD or pre-existing oxygen-dependent pulmonary diseases, severe broncho-pneumonia within 1 month prior to injury, steroid dependent asthma or uncontrolled asthma),
15. Pre-existing diseases which interfere with circulation (severe peripheral vascular disease, severe circulatory edema and/or lymphedema, regional lymph nodes dissection, significant varicose veins),
16. Any conditions that would preclude safe treatment or adding further risk to the basic acute burn trauma (such as a positive COVID test, severe immuno-compromising diseases, life threatening trauma, severe pre-existing coagulation disorder, severe cardiovascular disorder, significant pulmonary disorder, significant liver disorder including post alcoholic abuse impaired function or neoplastic disease, blast injury),
17. Chronic systemic steroid intake,
18. History of allergy and/or known sensitivity to pineapples, papaya, Bromelain or papain.
19. Enrollment in any investigational drug trial within 4 weeks prior to screening.

    -

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - University of South Alabama, Mobile, Alabama
  - Valleywise Health Medical Center, Phoenix, Arizona
  - University of California, Irvine, Orange, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Children's Hospital, University of Florida, Gainesville, Florida
  - University of Florida, Department of Surgery, Gainesville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Eskenazi Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Hospital, Kansas City, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins Bayview Medical Center, Burn Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Stony Brook University Medical Center, Stony Brook, New York
  - Akron Children's Hospital, Akron, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Legacy Oregon Burn Center, Portland, Oregon
  - Lehigh Valley Hospital and Health Network, Allentown, Pennsylvania
  - UPMC Mercy Burn Center, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Parkland Health & Hospital System, Burn Center, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - Colombia St Mary's Hospital, Milwaukee, Wisconsin